CLINICAL TRIAL: NCT00609401
Title: A Randomized Open Label Multicenter Phase II Study of First Line Therapy With Sorafenib in Association With IL-2 vs Sorafenib Alone in Patients With Unresectable and/or Metastatic Renal Cell Carcinoma
Brief Title: Study Comparing Association Between Sorafenib and Interleukin-2 (IL-2) Versus Sorafenib in 1st Line Therapy in Advanced (Adv) Renal Cell Carcinoma (RCC)
Acronym: ROSORC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Trial in Medical Oncology (Other)
Responsible Party: Giuseppe Procopio, ITMO
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number 2006-003137-32; EudraCT number 2006-003137-32
Record Dates: First submitted 2008-01-11; First posted 2008-02-07 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Metastatic Disease; Renal Cell Carcinoma
Keywords: Sorafenib; RCC; Metastatic disease
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — Sorafenib; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sorafenib 400 bid + IL-2 3 MU per 5 day/week for 2 weeks every 4
  Interventions: Drug: Nexavar (Sorafenib); Drug: IL-2
- 2 (Experimental): Sorafenib 400 mg bid
  Interventions: Drug: Nexavar (Sorafenib)

INTERVENTIONS:
Drug: Nexavar (Sorafenib) — 400 mg bid
Drug: IL-2 — IL-2 3 MU per 5 day/week for 2 weeks every 4
  Arms: 1

SUMMARY:
The ROSORC trial is a randomized study comparing the efficacy of a new association (sorafenib and IL-2) versus the standard therapy (sorafenib) in patients affected by different histotypes of metastatic RCC. This study is a first line therapy for the advanced disease. The primary objective is the progression free survival (PFS) in the 2 arms of therapy and the secondary objective is the overall survival (OS) and the response rate (RR) and the safety profile of the combination compared to sorafenib alone.

DETAILED DESCRIPTION:
Patients will be allocated in 2 groups:

ARM A - Sorafenib 400 mg twice daily continuously and low dose of IL-2 administered s.c.

ARM B - Sorafenib alone at the same dosage used in the previous arm

The trial is stratified according to the MSKCC prognostic model (low intermediate high risk) and histology (Clear cell vs other histotypes). The main inclusion criteria are: cytohistological diagnosis of RCC, measurable disease as RECIST criteria, signed written informed consent, life expectancy of greater than 3 months.

The efficacy and safety analysis will be performed on an intent to treat population.

The anticipated median PFS time in the control arm is 6 months and we will expect an increase of 3 months in the experimental arm.

The sample size is 128 patients, 64 in each arm (1:1 randomization)

The study started in November 2006 and is a multicenter Italian trial.

ELIGIBILITY:
Inclusion Criteria:

* Cytohistological diagnosis of RCC
* Written informed consent
* Measurable disease according to RECIST criteria
* Age >= 18 years
* Karnofsky PS >= 60%
* Life expectancy of greater than 3 months

Exclusion Criteria:

* Prior medical treatment for metastatic RCC
* Brain metastasis or spinal cord compression
* Chronic treatment with corticosteroids
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
PFS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Istituto Tumori Milano; E. Aitini, MD, Study Director — Ospedale di Mantova; M. Bregni, MD, Study Director — Ospedale San Raffaele Milano; G. Conti, MD, Study Director — Urologia - Ospedale di Como; M. Maio, MD, Study Director — Immunologia Oncologica - Ospedale Le Scotte Siena; G. Fasola, MD, Study Director — Ospedale di Udine; V. Zagonel, MD, Study Director — Medicina Oncologica - Ospedale Fatebenefratelli - Roma; S. Cascinu, MD, Study Director — Ospedale di Ancona; G. Marini, MD, Study Director — Ospedale di Brescia; A. Ardizzoia, MD, Study Director — Ospedale di Monza; Sergio Ricci, Prof., Study Director — Oncologia Medica - Ospedale Santa Chiara Pisa; L. Cavanna, MD, Study Director — Oncologia Piacenza; M. Aglietta, MD, Study Director — Ospedale di Candiolo Torino; A. Bertolini, MD, Study Director — SOC Oncologia Medica Azienda Ospedaliera Valtellina; Sergio Bracarda, MD, Study Director — Oncologia Medica Ospedale di Perugia; L. ISA, MD, Study Director — A.O. Melegnano - Gorgonzola; S. Monfardini, MD, Study Director — Oncologia Ospedale di Padova; D. Amadori, MD, Study Director — IOR Ospedale di Forlì; C. Porta, MD, Study Director — Ospedale San Matteo Pavia
Locations (1):
- Istituto Tumori, Milan, Italy

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Procopio G, Verzoni E, Bracarda S, Ricci S, Sacco C, Ridolfi L, Porta C, Miceli R, Zilembo N, Bajetta E; Italian Trials in Medical Oncology (ITMO) group. Overall survival for sorafenib plus interleukin-2 compared with sorafenib alone in metastatic renal cell carcinoma (mRCC): final results of the ROSORC trial. Ann Oncol. 2013 Dec;24(12):2967-71. doi: 10.1093/annonc/mdt375. Epub 2013 Sep 24. PMID 24063860